CLINICAL TRIAL: NCT00516490
Title: GnRH Agonist Administration in the Luteal Phase of ICSI-ET Cycles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AH-47/07
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2007-08-15 (Estimated); Status verified 2007-08

CONDITIONS: Infertility
Keywords: GnRH agonist; IVF/ICSI outcome; luteal phase
MeSH Terms: conditions — Infertility | interventions — Triptorelin Pamoate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): GnRH agonist administration
  Interventions: Drug: triptorelin acetate
- 2 (Placebo Comparator): Sterile saline injection
  Interventions: Drug: Na Cl %0.9

INTERVENTIONS:
Drug: triptorelin acetate — Single dose of 0.1 mg triptorelin subcutaneous injection on the 3rd day after embryo transfer
  Other Names: Decapeptyl Ferring GmBH Kiel Germany
  Arms: 1
Drug: Na Cl %0.9 — 0.1 ml sterile saline subcutaneous injection on the 3rd day after embryo transfer
  Other Names: Isotonik NaCl %0.09 Eczacibasi-Baxter Istanbul Turkey
  Arms: 2

SUMMARY:
A single dose GnRH agonist administration in the luteal phase of assisted reproduction cycles was reported to increase pregnancy and birth rates. This study was done to evaluate the reproducibility of previous findings.

DETAILED DESCRIPTION:
GnRH agonist administration in the luteal phase was reported to beneficially affect clinical outcome of ICSI-ET cycles. This randomized controlled trial evaluates the effect of a single dose GnRH agonist administered in the luteal phase on the outcome of ICSI - ET cycles stimulated with the long GnRH agonist protocol. Women undergoing embryo transfer following controlled ovarian hyperstimulation with a long GnRH agonist protocol were included. In addition to routine luteal phase support with progesterone women were randomized to receive a single dose of GnRH agonist or placebo on the sixth day after ICSI.Ongoing pregnancy rate was the primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing embryo transfer following controlled ovarian hyperstimulation with a long GnRH agonist protocol, oocyte pick-up and ICSI.
* Embryo transfer performed on day 3.

Exclusion Criteria:

* Participation in another trial that was being conducted in our unit at the same time.
* Preimplantation genetic screening cycles.
* Day 5 embryo transfers.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 570 (Actual)
Dates: Start 2006-09; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate beyond 20 weeks

SECONDARY OUTCOMES:
Clinical pregnancy
Embryo implantation rate

CONTACTS AND LOCATIONS:
Overall Officials: Baris Ata, M.D., Principal Investigator — The Assisted Reproduction Unit of the American Hospital of Istanbul; Bulent Urman, M.D., Study Director — The Assisted Reproduction Unit of the American Hospital of Istanbul
Locations (1):
- Amerikan Hastanesi Tüp Bebek Merkezi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Tesarik J, Hazout A, Mendoza-Tesarik R, Mendoza N, Mendoza C. Beneficial effect of luteal-phase GnRH agonist administration on embryo implantation after ICSI in both GnRH agonist- and antagonist-treated ovarian stimulation cycles. Hum Reprod. 2006 Oct;21(10):2572-9. doi: 10.1093/humrep/del173. Epub 2006 Aug 22. PMID 16926261
- [Derived] Ata B, Yakin K, Balaban B, Urman B. GnRH agonist protocol administration in the luteal phase in ICSI-ET cycles stimulated with the long GnRH agonist protocol: a randomized, controlled double blind study. Hum Reprod. 2008 Mar;23(3):668-73. doi: 10.1093/humrep/dem421. Epub 2008 Jan 12. PMID 18192671